CLINICAL TRIAL: NCT01451606
Title: Evaluating Duloxetine's Analgesic Effectiveness in Chronic Pelvic Pain
Brief Title: Duloxetine for the Treatment of Chronic Pelvic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Adequate recruitment was not achieved in the time frame allowed.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Joel Greenspan, Professor and Chair, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00047688
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Pelvis Pain Chronic
Keywords: Chronic Pelvic Pain (CPP); Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Duloxetine Hydrochloride; Sugars

STUDY DESIGN:
Intervention Model Description: One group receiving active drug treatment and second group receiving an indistinguishable placebo pill.
Who Masked: Participant, Investigator
Masking Description: Study drug allocation was determined by University pharmacy, using a random allocation algorithm unknown by researchers or patients.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo pill (Placebo Comparator): A pill that looks like the active drug, but does not contain any active ingredients.
  Interventions: Drug: Placebo
- Duloxetine (Active Comparator): The drug, Duloxetine, is marketed under the trade name Cymbalta. It is a serotonergic and noradrenergic reuptake inhibitor (SNRI).
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — 30 mg dose once daily, administered orally for 1 week, 60 mg dose once daily, administered orally for 5 weeks, 30 mg dose once daily, administered orally for 1 week
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Placebo — To serve as placebo for duloxetine. Administration schedule same as for active drug.
  Other Names: Sugar pill
  Arms: Placebo pill

SUMMARY:
This study is examining the effectiveness of duloxetine as a treatment for chronic pelvic pain in women. Duloxetine is FDA approved for the treatment of other pain conditions, including fibromyalgia and diabetic neuropathy.

DETAILED DESCRIPTION:
Chronic pelvic pain in women can be caused by various pathologies, such as endometriosis, fibroids, and adhesions. Surgical treatment of the pathology often relieves the pain, but a significant number of women continue to have pain, even after visibly successful surgery. One model explored in this study is that in some cases of chronic pelvic pain, the central nervous system has changed in its processing of pain-related signals, requiring a therapy directed to the Central Nervous System (CNS) to effectively treat the pain. This model has been supported in studies of other chronic pain conditions, such as fibromyalgia and migraine. This study will seek to determine whether the analgesic effectiveness of duloxetine is related to the pain state of the individual.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal adult women, aged 18-50
* Have chronic pelvic pain, as defined by the American College of Obstetrics and Gynecology
* Able to read and speak English

Exclusion Criteria:

* Chronic Pelvic Pain (CPP) only presenting in low back or vulva, or only present during menstruation or vaginal intercourse
* Self-report or documentation that all CPP sites were attributed by a prior physician to Irritable Bowel Syndromd (IBS), Interstitial cystitis (IC)/painful bladder syndrome (PBS), urinary tract infection, urinary stones, inflammatory bowel disease (ulcerative colitis or Crohn's disease), cancer or shingles.
* Currently pregnant or lactating
* A primary psychiatric diagnosis of major depression or history of suicide attempt as assessed by medical history. Also, those who would be considered to have Major Depressive Disorder (MDD) on the basis of the Diagnostic and Statistical Manual IV (DSM-IV) criteria will excluded, as well as those selecting "3" or "4" on item #9 of the Beck Depression Inventory (BDI; suicidal ideation).
* A history of bipolar disorder
* A history of seizure disorders
* Orthostatic Hypertension
* Exclusions based on the effects of duloxetine:

  1. Known hypersensitivity to duloxetine or the inactive ingredients in Cymbalta;
  2. Treatment with an monoamine oxidase inhibitor (MAOI) within 14 days of randomization, or potential need to use an MAOI during the study or within 5 days of discontinuation of the drug;
  3. Treatment with cytochrome P450 enzyme inhibitors;
  4. Uncontrolled narrow-angle glaucoma;
  5. Concurrent use of thioridazine
  6. Renal Impairment (serum creatinine of 1.5 or greater)
  7. History of jaundice or hepatomegaly
  8. Hepatic Insufficiency (elevated aspartate transaminase (AST), alanine transaminase (ALT), bilirubin, or Alkaline Phosphatase), tested at the screening period, after the first week of study medication, and again at the midpoint of the study.
* Participants who are taking Selective serotonin reuptake inhibitors (SSRIs), Selective serotonin and norepinephrine reuptake inhibitors (SSNRIs), monoamine oxidase inhibitors (MAOIs), or tricyclics within 14 days of randomization will be excluded.
* Participants who currently meet DSM-IV diagnostic criteria for Alcohol Abuse or Dependence
* Weight exceeding 285 pounds
* Hyponatremia, as determined by blood test results

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2015-11-04 (Actual); Study Completion 2015-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Greenspan, Ph.D., Principal Investigator — University Of Maryland Dental School
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 2011 - Dec. 2015. Recruitment from medical clinic and through public advertisements.
Pre-assignment Details: In person visit to complete eligibility screening.
Period: Overall Study
Arm/Group | Placebo Pill | Duloxetine
Started | 16 | 18
Completed | 12 | 15
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Pill | Duloxetine | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 11 | 21
  White | 4 | 6 | 10
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change in Rating of Spontaneous Pelvic Pain (0 -10 Scale).
Description: The primary clinical efficacy measure is the change in spontaneous (non-evoked) pelvic pain from the baseline period to the end of treatment. This was assessed by using the 0-10 numerical pain ratings to derive the primary outcome variable of clinical pain intensity difference due to treatment. Larger values (greater changes in ratings) are better outcomes.
Time Frame: Baseline and 8 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo Pill | Duloxetine
Number analyzed (Participants) | 12 | 15
units on a scale | 5 [2 to 8] | 5 [3 to 6.5]
Statistical Analysis 1: Comparison: Placebo Pill vs Duloxetine; Test type: Superiority; p = 0.52, Wilcoxon (Mann-Whitney) — Note that sample size was well below our target, making this test very low power

2. Secondary Outcome: Change in Endometriosis Health Profile - 30 Subscale for Functional Limitations Due to Pain
Description: This is a questionnaire assessment of functional limitations due to clinical pain. The range of scores for this subscale is 0-44. The measure is the change in score from baseline to end of treatment period. A greater number (change in score) is a better outcome.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Pill | Duloxetine
Number analyzed (Participants) | 12 | 15
units on a scale | 21.58 (26.73) | 12.92 (22.68)
Statistical Analysis 1: Comparison: Placebo Pill vs Duloxetine; Test type: Superiority; p = 0.84, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were recorded for the duration of a participants time in the study, including 2 weeks after end of treatment. For the entire study, AEs were noted from July 2011 - Dec. 2015.
Arm/Group | Placebo Pill | Duloxetine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 9/12 | 13/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pill (N=12) | Duloxetine (N=15)
Headache (Nervous system disorders) | 5 (5) | 5 (12)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (11)
Sleepiness (Nervous system disorders) | 2 (2) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No